CLINICAL TRIAL: NCT06539949
Title: Investigation of Efficacy of the Tony Robbins Rapid Planning Method (RPM) on Life Productivity and Mood States - a Controlled Experimental Trial
Brief Title: Efficacy of the Tony Robbins Rapid Planning Method (RPM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081040
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Stress; Mood; Motivation; Well-Being, Psychological; Self Esteem
Keywords: Seminar; Life Coach
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Subjects in the experimental group (RPM Group) will be admitted to the Tony Robbins Rapid Planning Method (RPM) virtually at no cost. RPM™ , developed by Tony Robbins, is a new system of thinking that is purported to help you align your daily actions with your life's purpose. During RPM, Tony will coach participants how to implement these life strategies.
  Interventions: Behavioral: Rapid Planning Method (RPM)
- Control (Active Comparator): Subjects assigned to the control group, will not attend the event, but instead be required to regularly complete journaling involving a to-do-list of their weekly work tasks.
  Interventions: Behavioral: Journaling

INTERVENTIONS:
Behavioral: Rapid Planning Method (RPM) — RPM is a three day immersive seminar. Subjects will be exposed to a variety of mind-body exercises and psycho educational content including neural linguistic programming, designed to motivate, inspire, and improve the quality of people's lives.
  Arms: Experimental
Behavioral: Journaling — Subjects will be keeping a weekly to-do list.
  Arms: Control

SUMMARY:
This study will consist of an experimental group and a control group. Approximately 150 adult males and females from the ages of 19+ will take part in this study. Subjects will be divided into a Control and Experimental Group. Subjects for the control and experimental group will be recruited from our internal database of subjects who have previously shown interest in studies and from userinterviews. Subjects in the experimental group (RPM Group) will be admitted to the Tony Robbins Rapid Planning Method (RPM) virtually at no cost, while the subjects assigned to the control group, will not attend the event, but instead be required to regularly complete journaling involving a to-do-list of their weekly work tasks. Psychological assessment surveys will be taken before the event, and at 1 week (day 8-13), and 4 weeks (day 29-34) post intervention. The control group will take the psychological assessment before beginning journaling, and at 1 week (day 8-13), and 4 weeks (day 29-34) post intervention.

DETAILED DESCRIPTION:
For the journaling control group, subjects will be asked to write a weekly to-do-list at least once weekly at the beginning of the week. And at least read, or refer to their journal on a daily basis as direction for the work activities of the day.

The 3-day RPM (Rapid Planning Method) event by Tony Robbins involves online seminar based training sessions designed to enhance participants' productivity, goal-setting abilities, and time management skills. On the first day, subjects engage in virtual workshops focused on establishing clear, specific, and achievable goals through the RPM framework, which emphasizes purpose-driven planning. Day two consists of interactive virtual sessions where participants develop personalized action plans, incorporating Robbins' strategies for prioritizing and organizing tasks. Throughout the event, participants partake in motivational exercises aimed at increasing engagement, self-efficacy, and clarity of vision. The final day includes collaborative virtual activities where subjects practice RPM techniques in real-world scenarios, receive feedback, and refine their plans.

Psychological assessment surveys will be taken before the event, and at 1 week (day 8-13), and 4 weeks (day 29-34) post intervention. The control group will take the psychological assessment before beginning journaling, and at 1 week (day 8-13), and 4 weeks (day 29-34) post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19+
* Male and Female
* English literate
* Willing to sign the study informed consent form
* Experimental group: must participant in Tony Robbins Rapid Planning Method (RPM)
* Control group: must be willing to journal regularly

Exclusion Criteria:

* Excluded from the experimental group if you DO NOT participate in RPM
* Excluded from the control group if you DO participate in RPM, or any other Tony Robbins sponsored event during the study intervention

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Purpose in life test | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  The PIL test is a 20-item self-report attitudinal scale designed to measure the extent to which a respondent perceives a general sense of meaning and purpose in life or respectively suffers from an "existential vacuum". This test is the first and the most-studied questionnaire to measure perceived life purpose and meaning. It consists of 11 items which focus on the respondents' mood (e.g., item 1: I am usually completely bored, neutral, exuberant, enthusiastic), 3 items which address life goals (e.g., item 3: In life I have no goals or aims at all, neutral, very clear goals and aims), and 3 items which address meaning of life itself (e.g., item 4: My personal existence is utterly meaningless without purpose, neutral, very purposeful and meaningful).
Work Extrinsic and Intrinsic Motivation Scale (WEIMS) | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  is divided into three-item six subscales, which correspond to the six types of motivation (i.e., intrinsic motivation, integrated, identified, introjected and external regulations, and motivation). Participants will be asked to indicate on a Likert-type scale ranging from 1 (does not correspond at all) to 7 (corresponds exactly) the extent to which the items represent the reasons they are presently involved in their work.
Life and productivity test | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  these are 30 Likert scale questionnaires, measured on a scale of 1 to 10, with 1 meaning "strongly disagree", and 10 meaning "strongly agree". It consists of 5 items which focus on the respondents productivity, 3 items which focus on time management skills, 4 items which focus on emotions, 14 items which focus on engagement, and 4 items which focus on clarity of vision and purpose.

SECONDARY OUTCOMES:
PERMA Profiler | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  The scale measures five aspects of well-being defined by Martin Seligman, PERMA - positive emotion, engagement, relationships, meaning, and accomplishment, as well as negative emotion and health.
Rosenberg's Self esteem scale | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The scale is believed to be uni-dimensional. All items are answered using a 4-point Likert scale format ranging from strongly agree to strongly disagree.

OTHER OUTCOMES:
Generalize Anxiety Disorder (GAD-7) | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  a self report-based survey that assesses generalized anxiety disorder and severity on a 7-item scale. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Perceived Stress Scale (PSS-10) | Pre - Event, 1 week Post - Event, 1 Month Post - Event
  measures global perceived stress via self-report on a ten item scale. Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Total scores ranging from 0-13 would be considered low stress. Total scores ranging from 14-26 would be considered moderate stress. Total scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- The Applied Science and Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared